CLINICAL TRIAL: NCT01926158
Title: Denosumab in Enhancement of Bone Bonding of Hip Prosthesis in Postmenopausal Women: a Randomized, Double-blind, Placebo-controlled Study
Brief Title: Denosumab in Enhancement of Bone Bonding of Hip Prosthesis in Postmenopausal Women
Acronym: ProliaHip
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Turku University Hospital (Other Government)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: ISS 20109714; 2011-000628-14 (EudraCT Number)
Record Dates: First submitted 2013-08-16; First posted 2013-08-20 (Estimated); Last update posted 2018-04-30 (Actual); Status verified 2018-04

CONDITIONS: Hip Osteoarthritis
Keywords: Denosumab; Osteoporosis; Hip replacement; Osteoarthritis; Radiostereometric analysis (RSA); Dual energy X-ray absorptiometry (DXA)
MeSH Terms: conditions — Osteoarthritis, Hip; Osteoporosis; Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Denosumab (Experimental): Subcutaneous injection of denosumab 60 mg 4 weeks before surgery and 22 weeks after surgery
  Interventions: Drug: Denosumb
- Placebo (Placebo Comparator): Subcutaneous injection of placebo 4 weeks before surgery and 22 weeks after surgery
  Interventions: Drug: Placebo (for denosumab)

INTERVENTIONS:
Drug: Denosumb — Prefilled syringe of 1 mL denosumab solution
  Other Names: Brand name: Prolia
  Arms: Denosumab
Drug: Placebo (for denosumab)
  Other Names: Prefilled syringe of 1 mL placebo solution
  Arms: Placebo

SUMMARY:
This randomized clinical trial will evaluate the efficacy of an antiresorptive osteoporosis drug (denosumab) in prevention of periprosthetic bone loss and in promotion of implant osseointegration (bone bonding) in postmenopausal women after total hip replacement. The investigators assume that denosumab prevents periprosthetic bone loss and enhances bone bonding of the hip stem in postmenopausal women.

DETAILED DESCRIPTION:
This is a randomized, double-blind and placebo-controlled trial to evaluate the efficacy of denosumab on the biologic incorporation of cementless hip prosthesis. The study population consists of sixty-eight postmenopausal female patients, who are scheduled to have cementless total hip replacement (THA) for primary hip osteoarthritis. The patients will be randomly assigned to receive a subcutaneous injection of denosumab 60 mg or placebo four weeks before surgery and 22 weeks after surgery. The primary hypothesis is that denosumab is effective in preventing periprosthetic bone loss in the proximal femur as measured by DXA. The secondary hypothesis is that denosumab is effective in enhancement of bone bonding (osseointegration) of cementless femoral stems, as measured by model-based radiostereometric analysis.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women, age: ≥ 60 years to ≤ 85 years at randomization
* Degenerative primary hip osteoarthritis as the indication of hip replacement
* Signed informed consent

Exclusion Criteria:

* Presence of severe osteoporosis (T-score less than -4.0 and a previous fracture)
* Presence of Dorr C-type geometric change of the proximal femur
* Evidence of secondary osteoporosis
* Clinical or laboratory evidence of hepatic disease
* Laboratory evidence of hypocalcaemia
* Vitamin D deficiency (serum 25-OH(D) < 12 ng/mL)
* Disorders of parathyroid function
* Uncontrolled hyperthyroidism or hypothyroidism
* History of malignancy, radiotherapy or chemotherapy for malignancy (except basal cell carcinoma of the skin) within the last 5 years
* History of osteonecrosis of the jaw
* History of recent tooth extraction or other dental surgery and/or invasive dental work planned in the next 2 years
* Severe asthma or chronic obstructive pulmonary disease
* History of solid organ or bone marrow transplant
* Use within 12 months of drugs that affect bone metabolism such as ant-osteoporotic agents (including SERMS), estrogens, testosterone, and anti-epileptics:

  * Cumulative dose of 500 mg prednisone or equivalent within the last 6 months
  * Ever use of oral or iv bisphosphonates
  * Ever use of strontium ranelate or fluoride
* Use of the following medications:

  * chronic systemic ketoconazole
  * androgens
  * cinacalcet
  * aluminum
  * lithium
  * protease inhibitors
  * gonadotropin-releasing hormone agonists
* Rheumatoid arthritis or any other inflammatory arthritis
* History of skeletal disorder, such as Paget's disease or osteomalacia
* Alcohol abuse
* General

  * Mental, neurological or other conditions that may affect the ability to perform functional or clinical assessments required by the protocol
  * Subjects with known sensitivity or intolerance to any of the products to be administered (calcium and D-vitamin supplements, denosumab)
  * Subject will not be available for protocol-required study visits, to the best of the subject's and investigator's knowledge
  * Any other condition that, in the judgement of the investigator, may compromise the ability of the subject to give written informed consent and/or to comply with all required study procedures

Ages: 60 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2013-12 (Actual); Primary Completion 2017-02-04 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Periprosthetic bone mineral density (BMD) | 48 weeks
  Periprosthetic BMD of the proximal femur will be measured according to seven Gruen zones and compared with the baseline value

SECONDARY OUTCOMES:
Radiostereometric analysis (RSA) of prosthesis stem migration | 48 weeks
  The translatory and rotatory migration of the femoral stem will be measured by means of model-based RSA and compared with the position at the baseline

OTHER OUTCOMES:
Functional recovery | 48 weeks
  To investigate if the enhanced incorporation of hip prostheses in denosumab treated patients compared to placebo leads to faster functional recovery as measured by main parameters of gait analysis, pedometer evaluation of walking activity and patient reported outcome measures

CONTACTS AND LOCATIONS:
Overall Officials: Hannu T Aro, MD, PhD, Principal Investigator — Turku University Hospital
Locations (1):
- Turku University Hospital, Turku, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aro HT, Alm JJ, Moritz N, Makinen TJ, Lankinen P. Low BMD affects initial stability and delays stem osseointegration in cementless total hip arthroplasty in women: a 2-year RSA study of 39 patients. Acta Orthop. 2012 Apr;83(2):107-14. doi: 10.3109/17453674.2012.678798. Epub 2012 Apr 11. PMID 22489886
- [Background] Moritz N, Alm JJ, Lankinen P, Makinen TJ, Mattila K, Aro HT. Quality of intertrochanteric cancellous bone as predictor of femoral stem RSA migration in cementless total hip arthroplasty. J Biomech. 2011 Jan 11;44(2):221-7. doi: 10.1016/j.jbiomech.2010.10.012. Epub 2010 Nov 11. PMID 21074160
- [Background] Alm JJ, Makinen TJ, Lankinen P, Moritz N, Vahlberg T, Aro HT. Female patients with low systemic BMD are prone to bone loss in Gruen zone 7 after cementless total hip arthroplasty. Acta Orthop. 2009 Oct;80(5):531-7. doi: 10.3109/17453670903316801. PMID 19916684
- [Background] Makinen TJ, Alm JJ, Laine H, Svedstrom E, Aro HT. The incidence of osteopenia and osteoporosis in women with hip osteoarthritis scheduled for cementless total joint replacement. Bone. 2007 Apr;40(4):1041-7. doi: 10.1016/j.bone.2006.11.013. Epub 2007 Jan 17. PMID 17239668
- [Background] Makinen TJ, Koort JK, Mattila KT, Aro HT. Precision measurements of the RSA method using a phantom model of hip prosthesis. J Biomech. 2004 Apr;37(4):487-93. doi: 10.1016/j.jbiomech.2003.09.004. PMID 14996560
- [Result] Nazari-Farsani S, Finnila S, Moritz N, Mattila K, Alm JJ, Aro HT. Is Model-based Radiostereometric Analysis Suitable for Clinical Trials of a Cementless Tapered Wedge Femoral Stem? Clin Orthop Relat Res. 2016 Oct;474(10):2246-53. doi: 10.1007/s11999-016-4930-0. Epub 2016 Jun 22. PMID 27334320